CLINICAL TRIAL: NCT04257058
Title: Predicting Childhood Cancer Survivors' Transition Readiness & Transfer Outcomes (SURV Transfer Outcomes) (Administrative Supplement to R01CA218389)
Brief Title: Education Tools to Support Pediatric Survivor Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jordan Marchak, Associate Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00091839; R01CA218389 (NIH)
Record Dates: First submitted 2020-02-04; First posted 2020-02-05 (Actual); Results first posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Pediatric Cancer
Keywords: Behavioral study; Social study; Pediatric cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Electronic educational material (Experimental): Participants in the trial included young adult survivors of childhood cancer. Participants completed an online pre-test survey via REDCap. After the pre-test is completed, participants review electronic media in REDCap. Study staff confirmed review of material and scheduled a post-test survey to be competed in REDCap two weeks after material is reviewed.
  Interventions: Behavioral: Electronic educational material

INTERVENTIONS:
Behavioral: Electronic educational material — Electronic media via email

SUMMARY:
This study aims to evaluate the impact of electronic educational materials on adolescent and young adult (AYA) survivors' knowledge about late effects, perceived benefits, self-efficacy, and intentions to engage in lifelong survivor care.

DETAILED DESCRIPTION:
Despite increased risk for morbidity and mortality related to cancer treatment, over half of young adult survivors of childhood cancer do not engage in the recommended healthcare designed to detect late effects and secondary cancers. There is a scarcity of data on adherence to survivor-focused healthcare, particularly at the critical transition from pediatrics to adult care. In order to improve transition outcomes, the investigators need to create media to educate survivors about need for adherence to adult survivor healthcare.

This study aims to evaluate the impact of electronic educational materials on AYA survivors' knowledge about late effects, perceived benefits, self-efficacy, and intentions to engage in lifelong survivor care.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 18-25 years of age,
* Diagnosed with cancer at ≤ 18 years of age,
* ≥ 2 years since the last cancer treatment,
* seen at least once in the Aflac Cancer Survivor Program (CSP) in the past 2 years or transitioned out of the Aflac CSP to adult survivor care since 2013.

Exclusion Criteria:

* Patients will be excluded from participation in the study if the participant is non-English speaking.
* Young adult survivors who are cognitively impaired and unable to complete the questionnaires.
* Participants that do not consent to the recording of their interviews.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 89 (Actual)
Dates: Start 2022-06-07 (Actual); Primary Completion 2024-04-13 (Actual); Study Completion 2024-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordan Marchak, PhD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This study and the data presented below only refers to the young adult survivors and does not include parents. Parents were not enrolled in this study. "Participants" refer to young adult cancer survivors.
Period: Overall Study
Arm/Group | Electronic Educational Material
Started | 89
Completed | 58
Not Completed | 31
Not completed — Lost to Follow-up | 31

BASELINE CHARACTERISTICS:
Arm/Group | Electronic Educational Material
Number analyzed (Participants) | 89
Age, Continuous [Mean (Standard Deviation); unit: years] | 19.8 (1.2)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 41
  Male | 45
  Non-Binary | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26
  Not Hispanic or Latino | 63
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 20
  White | 56
  More than one race | 3
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 89

OUTCOME MEASURES:

1. Primary Outcome: Survivor Care Knowledge Scale
Description: Knowledge was assessed at baseline and 2 weeks post-intervention, with the Survivor Care Knowledge scale, that includes 15-item multiple-choice quiz to assess participants' knowledge of the content covered in the electronic educational materials previously provided. Total score ranges from 0-15. Higher score is associated with better outcome.
Time Frame: Baseline, 2 weeks post-intervention
Population: Total number of participants analyzed per time point include participants that completed the corresponding visit and the specific assessment for this study outcome.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Educational Material
Number analyzed (Participants) | 89
score on a scale
  Baseline | 10.6 (2.1)
  2 weeks post-intervention: number analyzed (Participants) | 58
  2 weeks post-intervention | 11.2 (2.3)

2. Secondary Outcome: Benefits for Survivor Care
Description: 5-item study adapted Champion Benefits Scale for Mammography Screening. Total score ranges from 5-25. Lower score equals fewer perceived benefits of survivor care.
Time Frame: Baseline, 2 weeks post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Educational Material
Number analyzed (Participants) | 89
score on a scale
  Baseline | 12.6 (1.9)
  2 weeks post-intervention: number analyzed (Participants) | 58
  2 weeks post-intervention | 12.9 (1.8)

3. Secondary Outcome: Barriers for Survivor Care
Description: 11-item study adapted Champion Barriers Scale for Mammography Screening. Total score ranges from 11-55. Lower score equals fewer perceived barriers to survivor care.
Time Frame: Baseline, 2 weeks post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Educational Material
Number analyzed (Participants) | 89
score on a scale
  Baseline | 20.2 (5.9)
  2 weeks post-intervention: number analyzed (Participants) | 58
  2 weeks post-intervention | 19.9 (5.3)

4. Secondary Outcome: Perceived Susceptibility for Late Effects
Description: 3-item study adapted Champion Susceptibility Scale for Mammography Screening. Total score ranges from 3-15. Lower score equals less susceptibility to late effects of treatment.
Time Frame: Baseline, 2 weeks post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Educational Material
Number analyzed (Participants) | 89
score on a scale
  Baseline | 9.7 (3.1)
  2 weeks post-intervention: number analyzed (Participants) | 58
  2 weeks post-intervention | 10.4 (2.7)

5. Secondary Outcome: Intentions for Survivor Care
Description: 2-item study adapted Ajzen's Theory of Planned Behavior- Intentions. Total score ranges from 2-14. Lower score equals greater intention to engage in long-term follow-up care.
Time Frame: Baseline, 2 weeks post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Electronic Educational Material
Number analyzed (Participants) | 89
score on a scale
  Baseline | 11.8 (3.4)
  2 weeks post-intervention: number analyzed (Participants) | 58
  2 weeks post-intervention | 11.4 (3.4)

6. Secondary Outcome: Change in Perceived Health Competence Scale (PHCS)
Description: 8-item Perceived Health Competence Scale (PHCS). Total score ranges from 8-40. Lower score equals lower perceived health competence.
Time Frame: Baseline, 2 weeks post-intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Self-efficacy: Participants in the trial included young adult survivors of childhood cancer. Participants completed an online pre-test survey via REDCap. After the pre-test is completed, participants review electronic media in REDCap. Study staff confirmed review of material and scheduled a post-test survey to be competed in REDCap two weeks after material is reviewed.
Arm/Group | Self-efficacy
Number analyzed (Participants) | 89
score on a scale
  Baseline | 28.7 (5.2)
  2 weeks post-intervention: number analyzed (Participants) | 58
  2 weeks post-intervention | 27.0 (5.6)

ADVERSE EVENTS:
Time Frame: Information on adverse events was collected beginning at the time of the intervention and continuing through the end of the study, at 2 weeks post-intervention.
Arm/Group | Electronic Educational Material
All-Cause Mortality (participants affected / at risk) | 0/89
Serious Adverse Events (participants affected / at risk) | 2/89
Other Adverse Events (participants affected / at risk) | 0/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Electronic Educational Material (N=89)
Stroke (Nervous system disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/58/NCT04257058/Prot_SAP_001.pdf
  • Informed Consent Form (2023-07-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT04257058/ICF_000.pdf